CLINICAL TRIAL: NCT05093088
Title: ChronoBrain: Effect of Circadian Rhythm on Brain NAD Measured by Phosphorus Magnetic Resonance Spectroscopy at 7 Tesla
Brief Title: Effect of Circadian Rhythm on Brain NAD Measured by Phosphorus Magnetic Resonance Spectroscopy at 7 Tesla
Acronym: ChronoBrain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Collaborators: Nestle Health Science (Industry)
Responsible Party: Principal Investigator, Lijing Xin, Research Staff Scientist, Ecole Polytechnique Fédérale de Lausanne
Other Study IDs: 2021-00907
Record Dates: First submitted 2021-10-11; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Circadian Rhythm
Keywords: Circadian Rhythm; NAD; MRS; Lactate; reward; risk-taking
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Discovery of the circadian clock first established a genetic basis for behavior, and our understanding of circadian rhythm (CIR) has since expanded to provide molecular insights into physiology and disease. Yet the challenge remains to translate these insights regarding the role of the CIR in cells and tissues into the clinic. Many mechanistic pre-clinical experiments have shown that the CIR is directly linked with the Nicotinamide Adenine Dinucleotide (NAD) levels and the NAD redox ratio and that the NAD oscillation amplitude is diminished during aging and in the model of neurological diseases. Human ex-vivo data have also shown that NAD oscillates over time in human red blood cells. While mounting evidence in model organisms illustrate the central role of brain NAD for maintaining energy homeostasis and the CIR, similar data in human are sparse. To date, no study has been reported in human on the effect of the CIR on brain NAD levels.

NAD is a vital cofactor involved in brain bioenergetics for metabolism and Adenosine Tri-Phosphate (ATP) production, the energy currency of the brain. NAD exists in an oxidized (NAD+) or reduced (NADH) form, with NAD+/NADH (the redox ratio) being an important determinant of cytosolic and mitochondrial metabolic homeostasis. Additionally, NAD+ is a key substrate for multiple NAD+-dependent enzymes and is consumed by at least four class of enzymes involved in genomic stability, mitochondrial homeostasis, adaptive stress responses, and cell survival, including Sirtuins. Modulation of subcellular NAD+ synthesis can regulate the timing of signaling pathways. Mammalian circadian rhythms are coordinated with metabolic activity through controlled expression of Nicotinamide phosphoribosyltransferase (NAMPT). Regulation of NAMPT, in turn, results in oscillating NAD+ levels. The rhythmic oscillation of NAD+ serves as a feedback 'timer' by modulating the activities of NAD+-dependent enzymes, including sirtuins, helping to establish the periodicity of the cycles. NAMPT oscillations also dictate mitochondrial NAD+ levels and coordinate cellular respiration with awake periods. In these cases, modulation of NAMPT levels drives the rise and fall of NAD+ concentrations that serve to limit the duration of Sirtuins activity.

Fine control of neurometabolism is necessary for brain function, because neuronal firing produces dynamic changes in local energy demand. The Astrocyte Neuron Lactate Shuttle Hypothesis (ANLS) provides one way of understanding how these changing needs are met. In this model, neuronal activity increases extracellular glutamate, which stimulates increased glucose uptake and glycolysis in astrocytes. Within astrocytes, lactate is produced from pyruvate in a reversible manner by the lactate dehydrogenase enzyme in the cytoplasm. This enzyme requires NAD as a co-factor and one NADH is converted to NAD+ when one pyruvate molecule is converted to lactate. The astrocytes then release this lactate, increasing its extracellular concentration. Important to the ANLS hypothesis, lactate can be used by nearby neurons as an energy source.

Furthermore, under the influence of the CIR regulation, the human psychological and physiological functions fluctuate with time during the day. This effect has been observed in many cognitive domains, as well as in risky decision-making and reward function.

The hypothesis is that brain NAD level is modulated by the CIR and that the NAD redox ratio should increase during the day. The primary objective of this project is to determine the brain NAD status in the morning and in the afternoon. Many pre-clinical results have suggested a diurnal effect on brain NAD, yet no clinical data is available.

In this study, NAD+ and NADH level of the occipital region will be determined by 31P-MR spectroscopy at 7 T. Total NAD (tNAD) and NAD redox ratio NAD+/NADH will be calculated as well. Measurement will be conducted in the morning in the fasted state (AM session) and in the mid-afternoon (PM session) 3 hours after the lunch intake. To confirm that the AM and PM measurements are done in two different circadian states, salivary cortisol will be measured. Simultaneous detection of other energy metabolites (e.g. lactate, PCr, ATP) will be acquired for exploratory analysis. To explore how the NAD status correlates with behavioral measures of reward activation, the automatic Balloon Analogue Risk Task (BART) test will be performed at the end of each AM and PM session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males with age between 18 and 40 years
* Body Mass Index (BMI) = weight (kg) / height (m)2 between 18.5 to 25 kg/m2
* Able to understand and to sign a written informed consent prior to the study
* Informed consent signed
* Normal or corrected-to-normal vision
* Completed the Morningness-Eveningness Questionnaire (MEQ - Appendix B) and obtained a score between 30 and 70.
* No consumption of any beverages or foods with caffeine such as coffee and tea, within 24 hours prior to and during the experiment
* No strenuous exercise the day before the experiment. No strenuous exercise on the day of the experiment.
* Completed the one-week sleeping diary over the week before the experiment (Appendix A) showing habitually good sleep, such as falling asleep no later than midnight, waking up no later than 8:00 AM, and regularly having 7-9 hours of sleep every night.

Exclusion Criteria:

* Having any metallic, electronic, magnetic, or mechanical implants, devices, or objects, for safety reason linked to magnetic field exposure:

  * Aneurysm clip(s)
  * Cardiac pacemaker
  * Implanted cardioverter defibrillator (ICD)
  * Electronic implant or device
  * Magnetically-activated implant or device
  * Neurostimulation system
  * Spinal cord stimulator
  * Cochlear implant or implanted hearing aid
  * Insulin or infusion pump
  * Implanted drug infusion device, like portacath® for instance
  * Any type of prosthesis or implant
  * Artificial or prosthetic limb
  * Any metallic fragment or foreign body
  * Hearing aid
  * Other implants
* Claustrophobia
* Inability to perform tasks
* Significant psychological disorders
* Performing shift work or trans-meridian travel within one month before the study initiation
* Use of medication or nutritional supplements known to affect the circadian system or the NAD levels, including NAD precursor supplements.
* Hearing disorders (for safety purpose the participant should be able to hear from the operators during MRS scans)
* Subject having a hierarchical link with the investigator or co-investigators.
* Subject does not want to be informed of fortuitous discovery that could have an effect on his health

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy males with age between 18 and 40 years
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in brain NAD (NAD+; NADH, NAD+/NADH) measured by 31P-MRS between the two time points | two time points: morning (8:00-10:00) and afternoon (15:00-17:00)

SECONDARY OUTCOMES:
Change in brain lactate and BART test between the two time points | two time points: morning (8:00-10:00) and afternoon (15:00-17:00)

OTHER OUTCOMES:
association between end-point and other brain metabolites determined by 31P- and 1H-MRS | two time points: morning (8:00-10:00) and afternoon (15:00-17:00)

CONTACTS AND LOCATIONS:
Overall Officials: Lijing Xin, PhD, Principal Investigator — CIBM Center for Biomedical Imaging, École polytechnique fédérale de Lausanne (EPFL)
Locations (1):
- Center for Biomedical Imaging, École polytechnique fédérale de Lausanne (EPFL), Lausanne, Canton of Vaud, Switzerland